CLINICAL TRIAL: NCT02479022
Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Insulin 320 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NN1957-4195; 2014-003918-92 (EudraCT Number); U1111-1161-6716 (Other: WHO)
Record Dates: First submitted 2015-06-19; First posted 2015-06-23 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Level 1-7 escalating doses (Experimental)
  Interventions: Drug: Insulin 320; Drug: insulin glargine; Drug: placebo

INTERVENTIONS:
Drug: Insulin 320 — Subjects will be randomised to receive a single dose of Insulin 320 orally, at 7 escalating dose levels from 300 nmol to 21600 nmol. Progression to next dose level will be based on a safety evaluation.
Drug: insulin glargine — As an open label active comparator, subjects will be randomised to receive a single dose of insulin glargine subcutaneously (s.c., under the skin), at all dose levels. The insulin glargine dose will be the same at all dose levels.
Drug: placebo — Subjects will be randomised to receive a single dose of placebo orally as a comparator Insulin 320, at all dose levels.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the safety, tolerability, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of insulin 320 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18-55 years (both inclusive) at the time of signing informed consent
* Body mass index 18.5-28.0 kg/m^2 (both inclusive)
* Subject who is considered to be healthy based on the medical history, physical examination, and the results of vital signs, electrocardiograms and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Previous participation in this trial. Participation is defined as signed informed consent
* Any disorder which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol
* Presence of clinically significant acute and chronic gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea) as judged by the investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | From the time of trial product administration and until 12 days after trial product administration

SECONDARY OUTCOMES:
Area under the serum insulin concentration-time curve | From 0 to 288 hours after a single dose (SD)
Area under the glucose infusion rate-time curve | From 0 to 24 hours after a single dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com